CLINICAL TRIAL: NCT07317830
Title: The Effects of Eight Weeks of Supplementation With Two Vitamin D₃ Formulations in Adults With Subclinical and Clinical Vitamin D Deficiency: A Randomized Controlled Superiority Pilot Trial
Brief Title: Effects of Different Vitamin D3 Formulations in Vitamin D-Deficient Adults
Acronym: AMORPH-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Health Sciences, Serbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 302-27-01
Record Dates: First submitted 2025-12-12; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental 1 (Experimental): 2,000 IU of active ingredient (powder) per day
  Interventions: Dietary Supplement: Experimental 1 (powdered supplement)
- Experimental 2 (Active Comparator): 2,000 IU of active ingredient (oil) per day
  Interventions: Dietary Supplement: Experimental 2 (oily supplement)

INTERVENTIONS:
Dietary Supplement: Experimental 1 (powdered supplement) — Active powdered ingredient (2,000 IU/d)
  Arms: Experimental 1
Dietary Supplement: Experimental 2 (oily supplement) — Active oily ingredient (2,000 IU/d)
  Arms: Experimental 2

SUMMARY:
This randomized controlled superiority pilot trial will evaluate the efficacy of two vitamin D3 formulations administered over eight weeks in adults with subclinical or clinical vitamin D deficiency. The study will compare changes in serum 25-hydroxyvitamin D concentrations between formulations, as well as the proportion of participants who will achieve vitamin D sufficiency. Both formulations are expected to improve vitamin D status, with the hypothesis that one formulation will demonstrate superior bioavailability, resulting in greater and faster increases in circulating 25-hydroxyvitamin D. The findings will provide preliminary evidence to inform formulation selection and dosing strategies for correcting vitamin D deficiency and will support the design of larger, confirmatory trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over
* Serum 25(OH)D < 75 nmol/L
* BMI 18.5 - 29.9 kg/m2
* Free of clinically significant acute disorders and severe chronic diseases
* No planned travel to high-UV destinations or tanning bed use during the trial
* Willing to avoid non-study vitamin D supplements
* Able to give written informed consent and comply with study visits
* Submitted informed consent

Exclusion Criteria:

* Pregnancy of breast feeding
* Underweight or obesity
* History of any dietary supplement use within 8 weeks before screening
* Medications that materially alter vitamin D metabolism or calcium balance
* Subjects with a history of medicine or alcohol abuse
* Abnormal values for lab clinical chemistry (> 2 SD)
* Unwillingness to return for follow-up analysis
* Participation in other clinical trials within 60 days prior to screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
25(OH)D | Change from baseline 25(OH)D at 8 weeks
  Serum levels of 25(OH)D

SECONDARY OUTCOMES:
Total calcium | Change from total calcium at 8 weeks
  Serum levels of total calcium
Ionized calcium | Change from ionized calcium at 8 weeks
  Serum levels of ionized calcium
Phosphorus | Change from phosphorus at 8 weeks
  Serum levels of phosphorus
Magnesium | Change from magnesium at 8 weeks
  Serum levels of magnesium

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Study Chair — University of California, Los Angeles
Locations (1):
- Center for Health Sciences, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in vitamin D. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Only qualified researchers with academic interest in vitamin D research

REFERENCES:
- [Background] Vieira EF, Souza S. Formulation Strategies for Improving the Stability and Bioavailability of Vitamin D-Fortified Beverages: A Review. Foods. 2022 Mar 16;11(6):847. doi: 10.3390/foods11060847. PMID 35327269
- [Background] Dalek P, Drabik D, Wolczanska H, Forys A, Jagas M, Jedruchniewicz N, Przybylo M, Witkiewicz W, Langner M. Bioavailability by design - Vitamin D3 liposomal delivery vehicles. Nanomedicine. 2022 Jul;43:102552. doi: 10.1016/j.nano.2022.102552. Epub 2022 Mar 26. PMID 35346834
- [Background] Borel P, Caillaud D, Cano NJ. Vitamin D bioavailability: state of the art. Crit Rev Food Sci Nutr. 2015;55(9):1193-205. doi: 10.1080/10408398.2012.688897. PMID 24915331